CLINICAL TRIAL: NCT01942148
Title: A Multicenter, Open-label, Long-term Safety Study of Aripiprazole (Initial Dose 2 mg/Day, Maintenance Dose 6-24 mg/Day, Maximum Dose 30 mg/Day) Orally Administered Over 52 Weeks in Patients Who Complete a Short-term Treatment Study of Aripiprazole in Pediatric Patients (Aged 13-17 Years) With Schizophrenia (031-09-003 Study)
Brief Title: A Long-term, Extended Treatment Study of Aripiprazole in Pediatric Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 031-09-004; JapicCTI-101147 (Other: JAPIC)
Record Dates: First submitted 2013-09-10; First posted 2013-09-13 (Estimated); Results first posted 2017-06-28 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-04

CONDITIONS: Schizophrenia
Keywords: Schizophrenia, Pediatric patients
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aripiprazole (Experimental): Aripiprazole (initial dose 2 mg/day, maintenance dose 6-24 mg/day, maximum dose 30 mg/day) orally administered over 52 weeks to subjects who complete the 031-09-003 study
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole
  Other Names: Abilify

SUMMARY:
The objective of this study is to investigate the safety and efficacy of aripiprazole (initial dose 2 mg/day, maintenance dose 6-24 mg/day, maximum dose 30 mg/day) orally administered over a period of 52 weeks in subjects who complete a short-term treatment study of pediatric patients (aged 13-17 years) with schizophrenia (031-09-003 study).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of schizophrenia (295.30, 295.10, 295.20, 295.90, 295.60), according to DSM-IV-TR
* Male and female patients aged 13-17 years
* Patients completing the 031-09-003 study
* Patients who, in addition to their legal guardian, provide written informed consent, having understood the details of this study
* Inpatient or outpatient status

Exclusion Criteria:

* Patients who have a diagnosis of any other disease except schizophrenia, according to DSM-IV-TR
* Patients who have been compulsorily admitted to hospital
* Patients with mental retardation
* Patients with thyroid disorder
* Patients who fall under a contraindication listed in the ABILIFY package insert
* Patients with a serious hepatic, renal, cardiac or hematopoietic disorder
* Patients with a history or a complication of organic brain disorder or convulsive disorder such as epilepsy
* Patients with a history or a complication of diabetes and patients who fall under any of the following: fasting blood glucose level ≧ 126 mg/dL, non-fasting blood glucose level ≧ 200 mg/dL, HbA1c ≧ 6.5%
* Patients with a history or a complication of suicide attempt, suicidal thought or self-harm
* Patients with a score of ≧2(mild) on PART1 evaluation of CGI-SS
* Patients with a history or a complication of malignant syndrome, tardive dyskinesia or paralytic ileus
* Patients in a state of physical exhaustion accompanied by such conditions as dehydration or malnutrition
* Patients with a history or a complication of water intoxication
* Patients with Parkinson's disease
* Pregnant women, parturient women, nursing women, women of childbearing potential who wish to become pregnant during this trial. However, women of childbearing potential who are practicing an appropriate method of contraception (refer to 8.6) and have a negative pregnancy test result are eligible for inclusion in this study.
* Study enrollment is otherwise judged to be inappropriate by the Investigator or Subinvestigator

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2010-08; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyoji Imaoka, Mr, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (8):
- Japan (8):
  - Chubu Region
  - Chugoku Region
  - Hokkaido Region
  - Kansai Region
  - Kanto Region
  - Kyushu Region
  - Shikoku Region
  - Tohoku Region

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aripiprazole
Started | 68
Completed | 41
Not Completed | 27
Not completed — Adverse Event | 4
Not completed — Lack of Efficacy | 2
Not completed — Physician Decision | 11
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 8
Not completed — Use of the prohibition medicine | 1

BASELINE CHARACTERISTICS:
Arm/Group | Aripiprazole
Number analyzed (Participants) | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 68
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.1 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 37
Region of Enrollment [Number; unit: participants]
  Japan | 68

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline at Final Assessment in Positive and Negative Syndrome Scale (PANSS) Total Score
Description: The Positive and Negative Syndrome Scale (PANSS) is a 30-item scale where each symptom is rated on a severity scale ranging from 1-7: 1 =Absent, 2 =Minimal, 3 =Mild, 4 =Moderate, 5 =Moderate severe, 6 =Severe, 7= Extreme. PANSS total score is calculated by adding score of 30 items, which ranges from 30-210. Higher scores indicate worse condition.
Time Frame: Basline and Week52
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aripiprazole
Number analyzed (Participants) | 68
units on a scale | -7.9 (28.2)

2. Secondary Outcome: Mean Change From Baseline at Final Assessment in Clinical Global Impression-Severity of Illness (CGI-S) Score
Description: The Clinical Global Impression-Severity of Illness (CGI-S) Score is a clinician rated scale which assesses how mentally ill the patient is at the time. Scores range from 0 to 7: 0 = Not assessed, 1= Normal, not at all ill, 2 =Borderline mentally ill, 3= Mildly ill, 4= Moderately ill, 5= Markedly ill, 6= Severely ill, 7= Among the most extremely ill patients. Higher scores indicate worse condition.
Time Frame: Basline and Week52
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aripiprazole
Number analyzed (Participants) | 68
units on a scale | -0.3 (1.1)

3. Secondary Outcome: Mean Change From Baseline at Final Assessment in Children's Global Assessment Score (CGAS)
Description: The Children's Global Assessment Score (CGAS) is a rating scale which measures psychological, social and school functioning for children aged 6-17. Scores range from 0 to 100, with higher scores indicating better condition.
Time Frame: Baseline and Week52
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aripiprazole
Number analyzed (Participants) | 68
units on a scale | 5.6 (19.8)

ADVERSE EVENTS:
Time Frame: From the start date of screening examination to date of the final examination
Arm/Group | Aripiprazole
Serious Adverse Events (participants affected / at risk) | 7/68
Other Adverse Events (participants affected / at risk) | 61/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aripiprazole (N=68)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Delusion (Psychiatric disorders) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1)
Schizophrenia (Psychiatric disorders) | 5 (5)
Suicidal ideation (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aripiprazole (N=68)
Dental caries (Gastrointestinal disorders) | 5 (5)
Nausea (Gastrointestinal disorders) | 12 (15)
Vomiting (Gastrointestinal disorders) | 11 (26)
Gastroenteritis (Infections and infestations) | 4 (4)
Influenza (Infections and infestations) | 4 (4)
Nasopharyngitis (Infections and infestations) | 31 (43)
Otitis externa (Infections and infestations) | 4 (4)
Excoriation (Injury, poisoning and procedural complications) | 4 (4)
Contusion (Injury, poisoning and procedural complications) | 5 (8)
Weight decreased (Investigations) | 4 (4)
Akathisia (Nervous system disorders) | 8 (10)
Weight increased (Investigations) | 8 (8)
Headache (Nervous system disorders) | 9 (10)
Somnolence (Nervous system disorders) | 14 (15)
Tremor (Nervous system disorders) | 6 (6)
Insomnia (Psychiatric disorders) | 5 (8)
Schizophrenia (Psychiatric disorders) | 6 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No